CLINICAL TRIAL: NCT05035368
Title: Ladarixin 400 mg Twice a Day as Adjunctive Therapy to Improve Insulin Sensitivity and Glucometabolic Outcomes in Overweight Insulin-resistant Type 1 Diabetic Patients
Brief Title: Ladarixin as Adjunctive Therapy to Improve Insulin Sensitivity and Glucometabolic Outcomes in Type 1 Diabetes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Dompé decided to withdraw LDX0121 following an internal re-planning and an extensive review of the study design.
  At the time of withdrawal, no site had been activated and the drug had not been sent to investigators. No patients had been enrolled.
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LDX0121
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2022-01

CONDITIONS: Type I Diabetes
Keywords: Type I diabetes; Insulin-resistance; Overweight
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Overweight | interventions — 2'-((4'-trifluoromethanesulfonyloxy)phenyl)-N-methanesulfonylpropionamide

STUDY DESIGN:
Intervention Model Description: This study is a randomized, placebo-controlled, double-blinded, 2-arm, 2-period crossover phase II trial using the CXCR1/CXCR2 chemokine receptor antagonist ladarixin versus placebo as adjunctive therapy to insulin to improve insulin sensitivity as well as glucometabolic outcomes in adult, insulin-requiring, overweight, IR T1D patients.
  This trial will randomize 38 male and female patients 21-65 years of age, inclusive, with established insulin requiring T1D and IR. After a 2:1 randomization into a treatment sequence (either ladarixin followed by placebo, or placebo followed by ladarixin, respectively), patients will be followed up for a maximum of 53 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The identity of the treatment will remain unknown to the patient, Investigator, site staff, CRO and Dompé's Development personnel until the study is unmasked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ladarixin - placebo (Experimental): In this arm the treatment sequence is ladarixin 400 mg twice-a-day, followed by placebo, as adjunctive therapy to insulin in overweight, IR, T1D patients.
  IMP will be administered for 24 weeks in each treatment period with a 21-day washout between the two periods. (Ladarixin 24 weeks, washout 21 days, Placebo 24 weeks).
  Interventions: Drug: Ladarixin; Other: Placebo
- Placebo - Ladarixin (Experimental): In this arm the treatment sequence is placebo followed by ladarixin 400 mg twice-a-day, as adjunctive therapy to insulin in overweight, IR, T1D patients.
  IMP will be administered for 24 weeks in each treatment period with a 21-day washout between the two periods. (Placebo 24 weeks, washout 21 days, Ladarixin 24 weeks).
  Interventions: Drug: Ladarixin; Other: Placebo

INTERVENTIONS:
Drug: Ladarixin — Ladarixin will be administered orally at the dose of 400 mg twice a day at about 12-hour interval (morning and evening).
  Other Names: LDX
Other: Placebo — Placebo is administered with the same schedule of Ladarixin.

SUMMARY:
Objectives Primary study objective: To determine whether orally-administered ladarixin versus placebo adjunctive therapy improves insulin sensitivity in overweight, insulin-resistant (IR) type 1 Diabetic (T1D) adult subjects.

Secondary study objectives: To determine whether orally-administered ladarixin versus placebo adjunctive therapy is safe and well-tolerated in overweight, IR T1D adult subjects.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, double-blinded, 2-arm, 2-period crossover phase II trial using the CXCR1/CXCR2 chemokine receptor antagonist ladarixin versus placebo as adjunctive therapy to insulin to improve insulin sensitivity as well as glucometabolic outcomes in adult, insulin-requiring, overweight, IR T1D patients.

This trial will randomize 38 male and female patients 21-65 years of age, inclusive, with established insulinrequiring T1D and IR. After a 2:1 randomization into a treatment sequence (either ladarixin followed by placebo, or placebo followed by ladarixin, respectively), patients will be followed up for a maximum of 53 weeks.

The study database will be locked when the last patient randomized has completed visit 9 (week 52/53) and data have been cleaned.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of autoimmune T1D as documented by positive T1D diabetes-related autoantibodies [the presence at diagnosis of at least one or more of - Insulin autoantibodies (IAA), Anti-GAD (GAD65), Anti-IA2 (IA2), Zinc Transporter 8 (ZnT8) must be documented from medical records or new laboratory measurement (not including IAA)];
2. age 21-65 years at the time of consent;
3. T1D duration =>5 years;
4. current insulin standard of care (ISOC), either use of an insulin pump or a stable dose level and dose frequency (i.e. established dose range that does not fluctuate beyond 1SD of the median over a period of the last two months prior to enrollment), multiple daily injections of insulin (at least 3 injections per day) for the last two months prior to enrollment, with no plans to switch the modality of insulin administration during the 4 months following screening (e.g., injection user switching to a pump, pump user switching to injections);
5. HbA1c between 7.5%-10.0%, inclusive, as per results of screening laboratory measurement;
6. evidence of IR based on a total daily insulin dose >0.8 U/kg/ day and/or a screening estimated glucose disposal rate (eGDR) < 9 mg/kg/min 1-3 value strongly indicative of IR, sex- and ageadjusted;
7. subject is overweight or obese with a BMI of between 25-40 kg/m2, inclusive;
8. ability to comply with all protocol procedures for the duration of the study, including scheduled follow-up visits and examinations, and willing to be contacted by clinical trial staff;
9. provision of written informed consent prior of any study-related procedure not part of standard medical care.

Exclusion Criteria:

1. patients with known or suspected hypersensitivity to non-steroidal anti-inflammatory drugs or any excipient of the investigational medicinal products (e.g. lactose and croscarmellose) as well as patients with congenital lactase deficiency, galactosaemia or glucose-galactose intolerance will have to be excluded;
2. use of non-insulin medications for adjunctive blood glucose control (e.g: antidiabetic agents such as metformin, sulfonylureas, glinides, thiazolidinediones, exenatide, liraglutide, DPP-IV inhibitors, SGLT-2 inhibitors or amylin);
3. use of medications for weight reduction (such as: Belviq (lorcaserin), Qsymia (Phentermine + topiramate), Orlistat (xenical));
4. use of a medication such as stimulants, antidepressants and/or psychotropic agents that could affect weight gain or glycemic control of T1D;
5. subject is on treatment with drugs metabolized by CYP2C9 with a narrow therapeutic index [i.e., phenytoin, warfarin, and high dose of amitriptyline (>50 mg/day)];
6. any medications known to influence glucose tolerance (e.g. beta-blockers, angiotensin-converting enzyme inhibitors, interferons, quinidine antimalarial drugs, lithium, niacin, etc.);
7. evidence of cardiac QTcF > 470 msec and/or any history of significant cardiovascular disease/abnormality;
8. any condition, including unstable dietary approach and disordered eating behaviour patterns, that in the judgment of the investigator will adversely affect patient's safety or the completion of the protocol or otherwise confound study outcome;
9. pregnancy (females) based on serum test (quantitative beta hCG) at screening; unwillingness to use effective contraceptive measures up to 2 months following trial discharge (females and males);effective contraceptive measures include a hormonal birth control (e.g. oral pills, long term injections, vaginal ring, patch); the intrauterine device (IUD); a double barrier method (e.g. condom or diaphragm plus spermicide foam).
10. clinical diagnosis of celiac disease that is in poor control as defined by most recent tissue transglutaminase (tTG) that is in the abnormal range;
11. history of ≥1 Diabetic Ketoacidosis (DKA) events in the past 6 months;
12. history of ≥1 severe hypoglycemic events (cognitive impairment that required assistance to treat) in the past 6 months;
13. hypoalbuminemia defined as serum albumin < 3 g/dL ;
14. hepatic dysfunction defined by increased ALT/AST > 3 x upper limit of normal (ULN) and increased total bilirubin > 3 mg/dL [>51.3 μmol/L];
15. moderate to severe renal impairment calculated by estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.73 m2 as determined using Chronic Kidney Disease Epidemiology Collaboration (CKDEPI) creatinine equation;
16. poor accessibility to veins for blood collection;
17. past (within 1 month prior to randomization) or current administration of any immunosuppressive medications (including oral, inhaled or systemically injected steroids) and use of any investigational agents, including any agents that impact the immune response or the cytokine system;
18. condition which interferes with the ability to accurately determine glycated HbA1c. Examples include: Genetic variants (e.g. HbS trait, HbC trait), elevated fetal hemoglobin (HbF) and chemically modified derivatives of hemoglobin (e.g. carbamylated Hb in patients with renal failure); Any condition that shortens erythrocyte survival or decreases mean erythrocyte age (e.g., recovery from acute blood loss, hemolytic anemia); Iron deficiency anemia, iron replacement therapy;
19. significant systemic infection during the 4 weeks before the first dose of study drug (e.g., infection requiring hospitalization, major surgery, or i.v. antibiotics to resolve; other infections, e.g., bronchitis, sinusitis, localized cellulitis, candidiasis, or urinary tract infections, must be assessed on a case-bycase basis by the investigator regarding whether they are serious enough to warrant exclusion).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
The mean difference in glucose infusion rate (GIR) from baseline | Week 25 of each treatment period (visits 4 and 8)
  The glucose infusion rate (GIR) is a measure of the rate at which the patient receives intravenous administration of dextrose, which increases blood sugar levels. GIR is expressed in mg per kilogram body weight per minute (mg/Kg/min).

SECONDARY OUTCOMES:
Change from baseline of HbA1c levels | Week 25/26 (no later than 10 days after the last IMP dose) of each treatment period (visits 5 and 9)
  In this study glycated hemoglobin (HbA1c) must be between 7.5%-10.0%, inclusive, as per results of screening laboratory measurement.
Change in average (previous 3 days) daily insulin requirements | Week 25/26 (no later than 10 days after the last IMP dose) of each treatment period (visits 5 and 9)
  In this study insulin requirement is calculated as IU/kg/day averaged over the previous 3 days.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Giannoukakis, PhD, Principal Investigator — Allegheny General Hospital and West-Penn Hospital
Locations (1):
- Institute of Cellular Therapeutics Allegheny Health Network, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No